CLINICAL TRIAL: NCT06859866
Title: Efficacy of Adjunctive At-Home Photodynamic Therapy (aPDT) in the Treatment of Peri-Implant Mucositis: A Post-Marketing Interventional Pilot Study With a Medical Device
Brief Title: Efficacy of Adjunctive At-Home Photodynamic Therapy (aPDT) in the Treatment of Peri-Implant Mucositis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koite Health Oy (Industry)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PhoPIM
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Peri-implant Mucositis
Keywords: APDT; aMMP-8; antibacterial

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either the non-surgical treatment (TNC) group or the non-surgical treatment + Lumoral® (TNCL group) using sealed envelopes, with an equal number of envelopes for each treatment group. Each group will consist of 15 patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNC group (Active Comparator): Standard oral hygiene.
  Interventions: Other: Standard oral hygiene
- TNCL group (Experimental): Home-use antibacterial medical device.
  Interventions: Other: Standard oral hygiene; Device: The addition of home-based dual-light photodynamic therapy (Lumorinse® + Lumoral®)

INTERVENTIONS:
Other: Standard oral hygiene — Standard protocol includes oral hygiene instructions (OHI), professional supragingival and subgingival instrumentation, and air polishing. A combination of manual tools (scalers/curettes) and electric tools (sonic/ultrasonic instruments) will be used to remove plaque and tartar, with particular attention to avoid damaging the implant surface. Both supragingival and subgingival surfaces will be treated with the air polishing device using glycine powder. A local antiseptic (1% chlorhexidine gel) will be prescribed twice daily for 7 days after TNC. OHI will be reinforced at each follow-up visit.
Device: The addition of home-based dual-light photodynamic therapy (Lumorinse® + Lumoral®) — Lumorinse® is an effervescent tablet that provides a final concentration of indocyanine green (ICG) of 250 μg/mL when dissolved in 30 mL of water. After rinsing the mouth for 1 minute, the Lumoral® device is used to activate the ICG. The device consists of 48 LED lights in the shape of a mouthguard, which simultaneously provide antibacterial blue light (aBL) at 405 nm and near-infrared (NIR) LED light at 810 nm. In combination with the ICG photosensitizer, the device delivers simultaneous aBL and aPDT action on dental plaque. After 10 minutes of use (30 J/cm2 radiant exposure), the device automatically shuts off. After treatment, patients will follow regular home oral hygiene procedures according to the OHI provided.
  Arms: TNCL group

SUMMARY:
The study aims to establish a validated protocol enabling an alternative approach for bacterial biofilm control through the application of a novel at-home photodynamic/antibacterial blue light therapy in addition to non-surgical professional treatment (NST) for peri-implant mucositis. The primary outcomes will include reductions in plaque and bleeding scores, decreases in probing pocket depth, and lower aMMP-8 levels in PISF. Secondary outcomes will include changes in keratinized peri-implant mucosa (KPIM) and patient-reported outcome measures (PROMs).

DETAILED DESCRIPTION:
Dental implants offer an opportunity to restore oral health by replacing missing teeth, demonstrating exceptional longevity when properly maintained. The maintenance of implant health primarily depends on the effective removal of dental plaque, which is the primary cause of periodontal diseases, from both dental and prosthetic surfaces.

According to an accepted definition, peri-implant mucositis is an inflammation of the peri-implant mucosa without loss of supporting bone tissue, while peri-implantitis is characterized by inflammation of the peri-implant mucosa associated with supporting bone loss. Recent data indicate that a significant proportion, ranging from 50% to 90%, of implants are affected by peri-implant mucositis.

The diagnosis of peri-implant mucositis is currently based on clinical observations; however, clinical evaluations may yield false positives or fail to allow early diagnosis and timely treatment of pathological conditions. With the knowledge of the current restrictions, this study aims to evaluate the levels of active matrix metalloproteinase-8 (aMMP-8) derived from Peri-Implant Sulcular Fluid (PISF), which is one of the most precise and sensitive diagnostic markers of peri-implant tissue inflammation.

The treatment of peri-implant mucositis currently encompasses a range of professional and at-home measures. Typically, peri-implant mucositis precedes the characteristic bone loss of peri-implantitis; therefore, the timely treatment of clinical signs of inflammation is critical to prevent disease progression that could culminate in implant failure. Inadequate plaque removal increases the risk of peri-implantitis by hindering access to implant sites for oral hygiene, resulting in a higher incidence in areas that patients are unable to clean effectively compared to easily accessible sites, underscoring the importance of focusing on at-home dental care.

New methods for at-home oral care are under development, such as antimicrobial photodynamic therapy (aPDT), which utilizes a photosensitizer (PS) and low-intensity visible light to generate reactive oxygen species (ROS) that target pathogenic bacteria. Antibacterial blue light takes advantage of the intrinsic antimicrobial properties derived from endogenous photosensitizing chromophores of pathogenic microbes, eliminating the need for exogenous dyes.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 20 teeth within the oral cavity.
* Diagnosis of peri-implant mucositis: bleeding or suppuration upon gentle probing with or without increased probing depth compared to previous evaluations, and no bone loss beyond the changes in the crestal bone level resulting from initial bone remodeling.
* Patients willing and able to provide written informed consent.

Exclusion Criteria:

* Pregnancy.
* Patients with a history of periodontitis.
* Use of medications that could affect soft tissues within the past 6 months (e.g., antibiotics, anti-inflammatories, anticonvulsants, immunosuppressants, or calcium channel blockers, including doxycycline and bisphosphonates).
* Allergy to the photosensitizer.
* Patients with removable major prostheses or orthodontic appliances.
* Patients with untreated carious lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | 12 months
  Change in the inflammatory parameter BOP.A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual). Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus. Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent". BOP is reported as the percentage (%) of sites with positive findings.
  Calculation formula: number of bleeding sites/ 6 times number of teeth.
Bleeding on probing (BOP) | 6 months
  Change in the inflammatory parameter BOP.A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual). Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus. Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent". BOP is reported as the percentage (%) of sites with positive findings.
  Calculation formula: number of bleeding sites/ 6 times number of teeth.

SECONDARY OUTCOMES:
Visual Plaque Index (VPI) | 12 months
  Assessment of six index teeth, measured at four sites per tooth
  Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent" VPI reported as the percentage (%) of sites with plaque Calculation formula: number of sites with plaque/ 4 times number of teeth
Visual Plaque Index (VPI) | 6 months
  Assessment of six index teeth, measured at four sites per tooth
  Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent" VPI reported as the percentage (%) of sites with plaque Calculation formula: number of sites with plaque/ 4 times number of teeth
Peridontal Pocket Depth (PPD) | 12 months
  A full-mouth assessment, measured at six sites per tooth. Assessed from the base of the pocket to the gingival margin (mm)
Peridontal Pocket Depth (PPD) | 6 months
  A full-mouth assessment, measured at six sites per tooth. Assessed from the base of the pocket to the gingival margin (mm)
KIPM (Keratinized Implant Peri-implant Mucosa Width) | 12 months
  KMW is calculated at the midfacial as the distance in millimeters from the free mucosal margin to the mucogingival junction and classified as adequate (≥2 mm) or inadequate (<2 mm)
KIPM (Keratinized Implant Peri-implant Mucosa Width) | 6 months
  KMW is calculated at the midfacial as the distance in millimeters from the free mucosal margin to the mucogingival junction and classified as adequate (≥2 mm) or inadequate (<2 mm)
Biomolecular Analysis | 12 months
  The concentration of active Metalloproteinase-8 (aMMP-8) in peri-implant sulcular fluid (PISF) will be assessed with an ELISA test.
Biomolecular Analysis | 6 months
  The concentration of active Metalloproteinase-8 (aMMP-8) in peri-implant sulcular fluid (PISF) will be assessed with an ELISA test.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto De Biase, Professor, Principal Investigator — Department of Oral and Maxillofacial Sciences, Sapienza Università di Roma,
Locations (1):
- Department of Oral and Maxillofacial Sciences, Sapienza Università di Roma,, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nikinmaa S, Podonyi A, Raivio P, Meurman J, Sorsa T, Rantala J, Kankuri E, Tauriainen T, Patila T. Daily Administered Dual-Light Photodynamic Therapy Provides a Sustained Antibacterial Effect on Staphylococcus aureus. Antibiotics (Basel). 2021 Oct 13;10(10):1240. doi: 10.3390/antibiotics10101240. PMID 34680821
- [Background] Nikinmaa S, Alapulli H, Auvinen P, Vaara M, Rantala J, Kankuri E, Sorsa T, Meurman J, Patila T. Dual-light photodynamic therapy administered daily provides a sustained antibacterial effect on biofilm and prevents Streptococcus mutans adaptation. PLoS One. 2020 May 6;15(5):e0232775. doi: 10.1371/journal.pone.0232775. eCollection 2020. PMID 32374766
- [Background] Levine JI. Medications that increase photosensitivity. FDA document Dec 1990.
- [Background] Gomes SC, Romagna R, Rossi V, Corvello PC, Angst PD. Supragingival treatment as an aid to reduce subgingival needs: a 450-day investigation. Braz Oral Res. 2014;28. doi: 10.1590/S1806-83242014.50000004. PMID 25000595
- [Background] Alaijah, F., Morsi, A., Nasher, R. et al. Photobiomodulation therapy in the treatment of periodontal disease: a literature review. Laser Dent Sci 3, 147-153 (2019)
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Lahteenmaki H, Patila T, Raisanen IT, Kankuri E, Tervahartiala T, Sorsa T. Repeated Home-Applied Dual-Light Antibacterial Photodynamic Therapy Can Reduce Plaque Burden, Inflammation, and aMMP-8 in Peri-Implant Disease-A Pilot Study. Curr Issues Mol Biol. 2022 Mar 8;44(3):1273-1283. doi: 10.3390/cimb44030085. PMID 35723308
- [Background] Lang NP, Suvan JE, Tonetti MS. Risk factor assessment tools for the prevention of periodontitis progression a systematic review. J Clin Periodontol. 2015 Apr;42 Suppl 16:S59-70. doi: 10.1111/jcpe.12350. PMID 25496279
- [Background] Kassebaum NJ, Smith AGC, Bernabe E, Fleming TD, Reynolds AE, Vos T, Murray CJL, Marcenes W; GBD 2015 Oral Health Collaborators. Global, Regional, and National Prevalence, Incidence, and Disability-Adjusted Life Years for Oral Conditions for 195 Countries, 1990-2015: A Systematic Analysis for the Global Burden of Diseases, Injuries, and Risk Factors. J Dent Res. 2017 Apr;96(4):380-387. doi: 10.1177/0022034517693566. PMID 28792274
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of severe periodontitis in 1990-2010: a systematic review and meta-regression. J Dent Res. 2014 Nov;93(11):1045-53. doi: 10.1177/0022034514552491. Epub 2014 Sep 26. PMID 25261053
- [Background] Jepsen S, Berglundh T, Genco R, Aass AM, Demirel K, Derks J, Figuero E, Giovannoli JL, Goldstein M, Lambert F, Ortiz-Vigon A, Polyzois I, Salvi GE, Schwarz F, Serino G, Tomasi C, Zitzmann NU. Primary prevention of peri-implantitis: managing peri-implant mucositis. J Clin Periodontol. 2015 Apr;42 Suppl 16:S152-7. doi: 10.1111/jcpe.12369. PMID 25626479
- [Background] Berglundh T, Jepsen S, Stadlinger B, Terheyden H. Peri-implantitis and its prevention. Clin Oral Implants Res. 2019 Feb;30(2):150-155. doi: 10.1111/clr.13401. Epub 2019 Feb 3. PMID 30636066
- See also: Pereira PAB, Aho VTE, Paulin L, et al., (2017) Oral and nasal microbiota in Parkinson's disease. Parkinsonism and Related Disorders 38: 61-67 — https://doi.org/10.1016/j.parkreldis.2017.02.026